CLINICAL TRIAL: NCT03363477
Title: Demonstration of Pharmacodynamic Equivalence of Enoxaparin Rovi (100-mg Subcutaneous Injection) to Clexane® (100-mg Subcutaneous Injection) in Healthy Volunteers
Brief Title: Study of Pharmacodynamic Equivalence of Enoxaparin Rovi to Clexane®, in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ROV-RO20-2015-01; 2015-003489-10 (EudraCT Number)
Record Dates: First submitted 2017-11-29; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: antithrombotic; heparin; anticoagulant; low molecular weight heparin; pharmacodynamic equivalence
MeSH Terms: interventions — Enoxaparin; enoxaparin sodium

STUDY DESIGN:
Intervention Model Description: single-dose, randomized, double-blind, 2-period, 2-sequence crossover study
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study will be double blinded in that the subjects and laboratories will be blinded. While the enoxaparin (manufactured by Rovi, Spain) and Clexane (manufactured by Sanofi, EU) solutions for SC injection may be identical in appearance, the prefilled syringes for both study drugs may not be identical. Therefore, the unblinded pharmacist will be responsible for dispensing the study drug in a manner consistent with maintaining the blind and a dedicated unblinded team member will perform study drug administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AB treatment sequence (Experimental): Period 1-Test Treatment A: enoxaparin (100 mg/mL) 100-mg SC injection, manufactured by Rovi (Spain) Period 2-Reference Treatment B: Clexane (100 mg/mL) 100-mg SC injection, manufactured by Sanofi (EU)
  Interventions: Drug: Enoxaparin; Drug: Clexane
- BA treatment sequence (Active Comparator): Period 1-Reference Treatment B: Clexane (100 mg/mL) 100-mg SC injection, manufactured by Sanofi (EU) Period 2-Test Treatment A: enoxaparin (100 mg/mL) 100-mg SC injection, manufactured by Rovi (Spain)
  Interventions: Drug: Enoxaparin; Drug: Clexane

INTERVENTIONS:
Drug: Enoxaparin
  Other Names: Enoxaparin (Rovi, Spain); enoxaparin sodium
Drug: Clexane
  Other Names: Clexane (Sanofi, EU); enoxaparin sodium

SUMMARY:
To demonstrate the pharmacodynamic (PD) equivalence of enoxaparin Rovi (100 mg/mL) 100-mg SC injection to Clexane® (100 mg/mL) 100-mg SC injection in healthy volunteers.

As secondary objective, to evaluate the safety and tolerability of enoxaparin Rovi (100 mg/mL) in healthy volunteers.

DETAILED DESCRIPTION:
This is a single-dose, randomized, double-blind, 2-period, 2 sequence crossover study. Subjects will be screened up to 30 days before the study begins and admitted to the clinic on Day -1 of Period 1 for baseline assessments. Before dosing on Day 1 of Period 1, subjects will be randomly assigned to a treatment sequence. Subjects will receive a single dose of study drug on Day 1 of each treatment period.

On Day 1 of Period 1, subjects will receive a single dose by subcutaneous route of the assigned study drug: enoxaparin (100 mg/mL) 100-mg SC injection manufactured by Rovi Spain, or Clexane (100 mg/mL) 100-mg SC injection manufactured by Sanofi EU; after an overnight fasting period of at least 10 hours. Subjects will continue fasting for at least 4 hours after study drug administration.

The washout period between administrations of study drug in each period will be at least 7 days.

On Day 1 of Period 2, subjects will cross over to receive the dose of the other drug, after an overnight fasting period of at least 10 hours. The total duration of the study will be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides informed consent (approved by an Independent Ethical Committee (IEC)) before any study specific evaluation is performed.
2. Subject is between the ages of 18 and 45 years, inclusive.
3. All female subjects must have a negative pregnancy test at Screening and upon check-in to the clinic.
4. Women of childbearing potential must use or have used one of the following acceptable birth control methods: Surgical sterilization (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) for at least 6 months before the first dose of study drug;Intrauterine device in place for at least 3 months before the first dose of study drug; or barrier method (condom, diaphragm) for at least 21 days before the first dose of study drug and throughout the study.
5. Subject has a body mass index between 18 and 30 kg/m2, inclusive.
6. Subject is able and willing to abstain from alcohol from 48 hours before the first dose of study drug through the end of the study.
7. Subject has no clinically significant abnormalities in medical history, vital sign measurements, or physical examination findings.
8. Subject has computerized 12-lead electrocardiogram (ECG) results showing no signs of clinically relevant pathology or deviations, as judged by the investigator.
9. Subject has hematology, serum chemistry, coagulation, and urinalysis test results within the reference ranges (Hb ≥7.5 mmol/L and ≥8.5 mmol/L for female and male, respectively) or showing no clinically relevant deviations, as judged by the investigator. Thrombocytes at screening have to be within the normal range.
10. Subject is a nonsmoker or has quit smoking at least 6 months before the first dose of study drug.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria are met:

1. Subject has active or recurring clinically significant skin, head, ears, eyes, nose, throat, respiratory, cardiovascular, gastrointestinal, endocrine/metabolic, genitourinary, neurologic, hematologic, musculoskeletal, immunologic, allergic, psychological/psychiatric, or other disease requiring medical treatment.
2. Female subject with weight < 45 kg or male subject with weight < 57 kg.
3. Subject is a woman who is pregnant or breastfeeding.
4. Subject has systolic blood pressure greater than 150 mm Hg or diastolic blood pressure greater than 90 mm Hg at Screening (confirmed upon repeat measurement).
5. Subject has a calculated (Cockroft & Gault formula) creatinine clearance less than 80 mL/minute and the value does not return to within reference range upon retest.
6. Subject has Hb <7.5 mmol/L and <8.5 mmol/L for female and male, respectively.
7. Subject has an active malignancy of any type other than nonmelanomatous skin malignancies.
8. Subject has any history of alcohol abuse or drug addiction.
9. Subject has any history of relevant drug and/or food allergies.
10. Subject has used an investigational drug within 60 days before the first dose of study drug.
11. Subject has used any prescription drugs (with special attention to antiplatelet or anticoagulant medication, eg, acetyl salicylic acid, NSADs, clopidogrel, warfarin, acenocumarol, heparin, low molecular weight heparin, dabigatran, rivaroxaban, apixaban) or over-the-counter medication that may affect coagulation (including aspirin or NSAIDs) within 4 weeks before dosing, or any other over-the-counter medication (including vitamins, herbal supplements, or dietary supplements) within 2 weeks before dosing.
12. Subject has donated or lost 550 mL or more of blood (including plasmapheresis) within 60 days before the first dose of study drug.
13. Subject has a positive test result for drugs of abuse (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, oxycodone), cotinine, or alcohol.
14. Subject has a positive test result for human immunodeficiency virus (1 or 2) antibody, hepatitis B surface antigen, or hepatitis C virus antibody.
15. Subject has any illness within 5 days before the first dose of study drug.
16. Subject has a positive test for fecal occult blood at Screening.
17. Subject has any history and/or current conditions of bleeding tendency such as: active bleeding, known bleeding diathesis or hemostatic defects due to severe hepatic or renal disease; recent gastrointestinal or genitourinary bleeding (10 days before study entry) women of child-bearing potential with normal cyclic bleeding which is not considered as heavy menstruation by the investigator, are allowed for inclusion; diabetic hemorrhagic retinopathy, or other hemorrhagic ophthalmic conditions.
18. Subject has a known history or family history of any relevant congenital or acquired coagulation disorder (eg, hemophilia, von Willebrand-Jürgens syndrome, or activated protein C resistance based upon Factor V Leiden mutation).
19. Subject has a history of thrombocytopenia, including heparin induced thrombocytopenia.
20. Subject has a known history of hypersensitivity to drugs with a similar chemical structure to enoxaparin sodium (eg, unfractionated heparin, low molecular weight heparin) or to pork products.
21. Subject is a member of the professional or ancillary personnel involved in the study.
22. Subject is deemed not suitable for entry into the study in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
AUEC0-inf for anti-FXa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  area under the effect curve (AUEC) from time 0 to infinity, for anti-FXa
AUEC0-T for anti-FXa and anti-FIIa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  area under the effect curve (AUEC) from time 0 to the last measured activity (T), for anti-FXa and anti-FIIa
Amax for anti-FXa and anti-FIIa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  peak effect for anti-FXa activity (anti-FXamax), and anti-FIIa activity (anti-FIIamax)

SECONDARY OUTCOMES:
RAUEC | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  ratio of AUEC0-T of anti-FXa to anti-FIIa
Amax for TFPI levels | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  peak effect activity (Amax) forTissue factor pathway inhibitor (TFPI)
AUEC0-T for TFPI levels | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  Area under the effect curve (AUEC) from time 0 to the last measured activity (T) forTissue factor pathway inhibitor (TFPI)
AUEC0-inf for TFPI levels | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  Area under the effect curve (AUEC) from time 0 to infinity forTissue factor pathway inhibitor (TFPI)
Tmax for anti-FXa and anti-FIIa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  time of observed maximum measured plasma activity for anti-FXa and anti-FIIa
t1/2 for anti-FXa and anti-FIIa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  apparent first order terminal elimination half-life for anti-FXa and anti-FIIa
CL/F for anti-FXa and anti-FIIa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  apparent plasma clearance after extravascular administration for anti-FXa and anti-FIIa
MRT for anti-FXa and anti-FIIa | Day -1 (Periods 1 and 2), before dosing (Pre-dose), and between 0.5 and 36 hours after dosing on Day 1 (Periods 1 and 2)
  mean residence time for anti-FXa and anti-FIIa
Adverse Events (AEs) | from Informed Consent signature until 14 days after the last study drug administration (independently of the period)
  All treatment emergent AEs (TEAEs), relationship of TEAEs to study drug, severity of TEAEs, treatment emergent serious AEs, relationship of treatment emergent serious AEs to study drug, and TEAEs leading to study drug discontinuation. The frequency of TEAEs will be summarized by system organ class and preferred term
hematology | at Screening, Day -1 (Period 1 only), and Day 3 (Period 2 only) and at the follow up visit (Day 7 of Period 2 only)
  clinical laboratory results
Serum chemistry | at Screening, Day -1 (Period 1 only), and Day 3 (Period 2 only) and at the follow up visit (Day 7 of Period 2 only)
  measurements of a variety of compounds in the serum layer of blood
Coagulation | at Screening, Day -1 (Period 1 only), and Day 3 (Period 2 only) and at the follow up visit (Day 7 of Period 2 only)
  Prothrombin time (reported in seconds) and activated partial thromboplastin time (aPTT)
Urianalysis | at Screening, Day -1 (Period 1 only), and Day 3 (Period 2 only) and at the follow up visit (Day 7 of Period 2 only)
  measurements of a variety of compounds in urine
Blood presure | at Screening, Day -1 (Period 1 only), and before dosing (Pre-dose) and 0.5 hours after dosing on Day 1 (Periods 1 and 2)
  systolic and diastolic blood presure recorded after the subject had been resting for at least 5 minutes
Pulse rate | at Screening, Day -1 (Period 1 only), and before dosing (Pre-dose) and 0.5 hours after dosing on Day 1 (Periods 1 and 2)
  recorded after the subject had been resting
Respiratory rate | at Screening, Day -1 (Period 1 only), and before dosing (Pre-dose) and 0.5 hours after dosing on Day 1 (Periods 1 and 2)
  measured subsequently to pulse rate
Tympanic temperature | at Screening, Day -1 (Period 1 only), and before dosing (Pre-dose) and 0.5 hours after dosing on Day 1 (Periods 1 and 2)
  measured subsequently to pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: Maria Velinova, MD, PhD, Principal Investigator — PRA Health Sciences (PRA) - Early Development Services (EDS)

IPD SHARING:
Plan to Share IPD: No